CLINICAL TRIAL: NCT01597674
Title: A Double-blind, Placebo-controlled, Parallel-group Study of the Effect of 5, 10 and 25 mg Daily of YF476 for 14 Days on 24-hour Ambulatory Gastric pH and Plasma Gastrin Concentrations in Healthy Volunteers
Brief Title: Effect of 5, 10 or 25 mg of YF476 Daily for 14 Days on Stomach Acidity in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trio Medicines Ltd. (Industry)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 97-010
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Reflux Oesophagitis
Keywords: YF476; gastrin receptor antagonist; gastric pH; gastrin; healthy subjects
MeSH Terms: conditions — Esophagitis, Peptic | interventions — YF 476

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: YF476 — There were 4 treatments: 3 dose levels of YF476 (5mg, 10mg, 25 mg) and placebo.
  Each treatment taken by mouth once daily for 14 days (Study Days 1-14). Each subject took 1 of the 4 treatments.

SUMMARY:
The objective of the study was to assess whether the tolerance to the effect of YF476 on gastric pH observed with repeated doses in a previous study in healthy volunteers can be avoided by using smaller doses of YF476.

DETAILED DESCRIPTION:
YF476 is a novel, potent and selective gastrin antagonist that inhibits basal and meal-stimulated gastric acid secretion, enhances gastric emptying of a liquid meal and increases lower oesophageal sphincter pressure in animals. In a placebo- and ranitidine-controlled, crossover study in healthy volunteers, single doses of 5, 25 and 100mg of YF476 increased gastric pH; the effect was dose-dependent in magnitude and duration and compared favourably with that of ranitidine 150mg. In a placebo- and omeprazole-controlled, parallel-group study in healthy volunteers, 25 and 100mg of YF476 twice daily for 7 days, did not significantly affect gastric pH unlike omeprazole 20mg daily for 7 days. YF476 and omeprazole both increased plasma gastrin concentrations. Single and repeated doses of YF476 were well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-45 years.
* No clinically relevant abnormal findings in the clinical history or physical examination at the screening assessment which could interfere with the objectives of the study or make the subject's participation hazardous.
* No clinically relevant abnormal laboratory values at the screening evaluation (Attachment 2).
* A normal ECG at the screening examination.
* A body mass index (Quetelet index) in the range 19.0-30.9:

  *Body Mass Index = weight [kg]_ height [m]2
* Subjects must be of sufficient intelligence to understand the nature of the study and any hazards of their participation in it. They must be able to communicate satisfactorily with the Investigator and to participate in, and comply with the requirements of, the entire study.
* Subjects must give their written consent to participate after reading the Information-for-Volunteers Leaflet and Consent Form, and after having the opportunity to discuss the study with the Investigator or his deputy.

Exclusion Criteria:

* Clinically relevant abnormal history or physical findings at the screening assessment, which could interfere with the objectives of the study or the safety of the subject's participation.
* Clinically relevant abnormalities of laboratory values or ECG at screening evaluation.
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate subject's participation in the study or make it unnecessarily hazardous.
* Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease or history of any psychotic mental illness.
* Participation in other clinical studies of a new chemical entity or a prescription medicine within the previous 3 months.
* Presence or history of drug or alcohol abuse, or intake of more than 40 units of alcohol weekly.
* Loss of more than 400mL blood during the 3 months before the study, e.g. as a blood donor.
* Use of prescription medication during 30 days before the study.
* Use of an over-the-counter medicine during 7 days before the study
* Blood pressure and heart rate in seated position at the screening examination outside the ranges 90-150mmHg systolic, 40-90mmHg diastolic; heart rate 40-100 beats/min.
* Possibility that the subject will not cooperate with the requirements of the protocol.
* Evidence of drug abuse on urine testing at study entry.
* Positive test for hepatitis B or C or HIV 1 & 2.
* High risk of hepatitis or HIV infection.
* History of severe allergic disease.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 1997-04; Primary Completion 1997-06 (Actual); Study Completion 1997-06 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic parameters: gastric pH and plasma gastrin | 8 weeks
  On Study Days 1, 7 and 14, ambulatory gastric pH recorded continuously from 0.5h before dosing until 24h after dosing. Subjects dosed between 0900-0930h. Standard meals and a drink (decaffeinated) taken at 4, 9, 13 and 22 h after dosing. Water (150mL) given at 2, 6, 8 and 11 h after dosing.
  On Study Days 1, 7 and 14, blood samples (4mL) taken via a cannula for assay of plasma gastrin at 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 16, 18, 20, 22 and 24 h after dosing.
Clinically relevant changes from baseline in safety assessments | 8 weeks
  Physical examination, ECG and safety tests of blood/urine at screening and at follow up.
Numbers of adverse events | 8 weeks
  Adverse events throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Boyce, Study Director — Trio Medicines Limited
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom